CLINICAL TRIAL: NCT07281547
Title: Mechanistic Randomized Controlled Feasibility Trial of Aspirin on Endometrium and Inflammatory Metabolites in Postmenopausal Women With Non-Atrophic Endometrial Changes
Brief Title: Low Dose Aspirin to Lower Inflammation and Prevent Endometrial Cancer in Postmenopausal Women With Non-atrophic Endometrial Changes and Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MC240602; NCI-2025-08686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006515 (Other: Mayo Clinic Institutional Review Board); MC240602 (Other: Mayo Clinic)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Specimen Handling; Aspirin; Watchful Waiting; Observation; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (low dose aspirin) (Experimental): Participants receive low dose aspirin PO QD for up to 42 days in the absence of unacceptable toxicity. Additionally, patients undergo pelvic ultrasound and blood, urine, and endometrial tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Low-Dose Aspirin; Other: Questionnaire Administration; Procedure: Ultrasound Imaging
- Arm II (observation) (Active Comparator): Participants undergo observation for up to 42 days in the absence of unacceptable toxicity. Additionally, patients undergo pelvic ultrasound and blood, urine, and endometrial tissue sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Patient Observation; Other: Questionnaire Administration; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood, urine, and endometrial tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Low-Dose Aspirin — Given PO
  Other Names: Baby Aspirin
  Arms: Arm I (low dose aspirin)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm II (observation)
Other: Questionnaire Administration — Ancillary studies
Procedure: Ultrasound Imaging — Undergo pelvic ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase IV trial studies whether low dose aspirin can be used to lower inflammation and prevent endometrial cancer in postmenopausal women with changes in the endometrial tissue that are not related to thinning (non-atrophic endometrial changes) and pain. As people age, there is an accumulation of fats, cell death, and inflammation, which causes a surge of pro-cancer-causing events. It is thought that there are several factors involved in the development of endometrial cancer, but that managing the inflammation may address the root cause. Low dose aspirin is aspirin that contains a lower dose than a standard adult tablet. Aspirin is a drug that reduces pain, fever, inflammation, and blood clotting. Aspirin belongs to the family of drugs called nonsteroidal anti-inflammatory agents. It is also being studied in cancer prevention. Giving low dose aspirin may be an effective way to lower inflammation and prevent endometrial cancer in postmenopausal women with non-atrophic endometrial changes and pain.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Postmenopausal women
* PRE-REGISTRATION: Transvaginal ultrasound
* PRE-REGISTRATION: Scheduled endometrial biopsy
* PRE-REGISTRATION: Provide risk factor survey
* REGISTRATION: Postmenopausal (defined clinically by no period for over 1 year or postmenopausal follicle-stimulating hormone [FSH], estradiol, or anti-Mullerian hormone [AMH] levels due to natural, medical, or surgical causes)
* REGISTRATION: Have pain (an indicator of inflammation) and other findings warranting endometrial sampling (postmenopausal bleeding [PMB], incidentally noted thickened endometrium > 4mm on ultrasound, obesity, fibroids)
* REGISTRATION: Capable of providing informed consent
* REGISTRATION: Understands English or Spanish language for consent and questionnaires
* REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance
* REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research
* REGISTRATION: Willingness to provide mandatory urine sample for correlative research

Exclusion Criteria:

* PRE-REGISTRATION: Not postmenopausal person born with uterus
* PRE-REGISTRATION: Atrophic endometrium
* PRE-REGISTRATION: No uterus
* PRE-REGISTRATION: Malignancy found
* REGISTRATION: Patients with previous hysterectomy (removal of the uterus)
* REGISTRATION: Atrophic endometrium on endometrial sampling performed clinically
* REGISTRATION: Patients from outside the Mayo Clinic Comprehensive Cancer Center (MCCCC) area
* REGISTRATION: Clinically contraindicated to discontinue use of anticoagulation other than aspirin
* REGISTRATION: Contraindication to use of nonsteroidal anti-inflammatory drugs (NSAIDs) or previous adverse reaction or intolerance to NSAIDs
* REGISTRATION: History of uterine, cervical, or ovarian cancers or precancers (endometrial hyperplasia, cervical dysplasia, fallopian tube intraepithelial carcinoma)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-12-11 (Estimated); Study Completion 2028-12-11 (Estimated)

PRIMARY OUTCOMES:
Change in prostaglandin E2 (PGE2) | Baseline to 6 weeks
  Assessed by repeated tissue sampling of the endometrium and compared between treatment and observation groups. A linear mixed-effects model (LMM) will be used to compare the change in PGE2 levels obtained from paired endometrial sampling between two groups of patients (aspirin versus [vs.] no aspirin). The continuous time that elapses between sampling will be assessed together with the binary patient group (aspirin vs. no aspirin) to investigate the change in continuous PGE2 measurement.

SECONDARY OUTCOMES:
Facilitators and Barriers to Participating in a Clinical Trial After Consenting to Clinical Trial | Baseline to 6 weeks
  Assessed at baseline (after consent to participate) using a questionnaire developed for this study: Facilitators and Barriers to Participating in a Clinical Trial After Consenting to Clinical Trial. The survey consists of 7 questions evaluating motivation for participating, barriers to participating, and expectations and understanding of study outcomes. Questions can be answered with one of the listed multiple choice options or with an open-ended "other" option. Post-study data collection will be completed via interview using questions similar to the baseline survey. Results will be analyzed and reported descriptively.

OTHER OUTCOMES:
Correlation of biomarkers with endometrial status | Baseline to 42 days
  Biomarkers obtained from biospecimen samples will be assessed for correlation with endometrial status in women on low-dose aspirin versus those not taking low-dose aspirin (observational cohort). Biomarker data will be tested in LMMs for significant association with treatment group and change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. DeStephano, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials